CLINICAL TRIAL: NCT06090396
Title: Non-invasive Cardiac Index Monitoring in Young Children During the Perioperative Period: Quantitative Comparison of Electrical Cardiometry and Transthoracic Echocardiography
Brief Title: Non-invasive Cardiac Index in Children
Acronym: NICIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laszlo Vutskits (Other)
Responsible Party: Sponsor-Investigator, Laszlo Vutskits, Head of Paediatric Anaesthesia, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: GE 2023-00672
Record Dates: First submitted 2023-10-05; First posted 2023-10-19 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Output; Anesthesia; Infant ALL
Keywords: hemodynamics; electrical cariometry; non-invasive; infant
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cardiac output monitoring with electrical cardiometry — comparison of limits of agreement between the two monitoring modalities
  Other Names: cardiac output monitoring with transthoracic echocardiography

SUMMARY:
This study investigates the level of agreement of two non-invasive cardiac output monitors (transthoracic echocardiography and electrical cardiometry) in young children under anesthesia.

DETAILED DESCRIPTION:
Young children are particularly prone to hemodynamic instability during the perioperative period which, in turn, may lead to organ morbidity. Currently, in routine surgical procedures in otherwise healthy children, hemodynamic status in the perioperative period is primarily assessed by non-invasive systemic blood pressure management. While this approach can detect systemic arterial hypotension, it does not provide us with guidance on whether the decrease in blood pressure is the result of changes in cardiac output and/or in systemic vascular resistance. This information would be important to know since treatment modalities may differ.

Recent technical development in electrical cardiometry allows us to non-invasively monitor cardiac output. The accuracy of the method has been validated in neonatal and paediatric cohorts, and electrical cardiometry is now regularly used to monitor cardiac output in the perioperative setting. Nevertheless, the trending patterns of cardiac output in otherwise healthy young children undergoing routine surgical procedures, still need to be described. Due to technical aspects, transthoracic echocardiography is now recognised as "gold-standard" measurement of cardiac output in paediatric patients.

This study is based on a commonly and non-invasively applied monitoring equipment (ICON) which is now regularly used on anesthetized children for the detection of cardiac output during the perioperative period. The primary objective of this validation study is to confirm the non-inferiority of cardiac output measurement with electrical cardiometry versus transthoracic echocardiography in young children ( 0-17 months of age) during the perioperative period.

The secondary objective is to describe the trending aspects of cardiac output during the anaesthesia until the recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0 to 17 months included
2. Greater than 36 weeks post-menstrual age (PMA) on the day of the study
3. Undergoing general anaesthesia for surgery that is expected to last more than 30 minutes (combines anaesthesia and surgical time)
4. Parental/guardian understands and reads French and permission (informed consent) obtained
5. ASA 1-3 status

Exclusion Criteria:

1. Structural/anatomical anomaly or other circumstances (e.g., patient positioning) making it difficult to apply the sensors to the body or limiting the feasibility of the TTE
2. Any Congenital heart diseases
3. Known allergy to electrodes' glue
4. Thoracic, cardiac and head surgery
5. Traumatic surgery with hemodynamic instability

Ages: 0 Months to 17 Months | Sex: All
Age Groups: Child
Study Population: Project population: infants (ASA1-3 status) up to 18 months of age undergoing a surgical procedure under general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Cardiac output measured by transthoracic electocardiometry ICON®- expressed as L/minutes | During the intraoperative period, up to 30 minutes after anesthesia induction
  This parameter is widely used in validation studies aimed to assess cardiac output
Cardiac output measured by Transthoracic echocardiography - expressed as L/minutes | During the intraoperative period, up to 30 minutes after anesthesia induction
  This parameter is widely used in validation studies aimed to assess cardiac output
Estimation of bias between cardiac outputs measured by ICON and Transthoracic echocardiography | During the intraoperative period, up to 30 minutes after anesthesia induction
  This statistical description is widely used in studies comparing accuracy/agreement between two different measurement modalities using the same units of measurements; it does not have a physical unit of measure

SECONDARY OUTCOMES:
The secondary endpoints are the bias in the temporal trend of changes between ICON®- and TTE-derived cardiac index values, and the Mean Percentage Error (MPE). | During the intraoperative period, up to 30 minutes after anesthesia induction
  These are statistical parameters and they do not have a physical unit of measure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided